CLINICAL TRIAL: NCT03889405
Title: Clinical Study Evaluating the Safety of Invu ™ and Comparative Performance of Invu ™ Versus IUPC in Prenatal Monitoring of Pregnant Subjects With Uterine Contractions.
Brief Title: Comparative Performance of INVU™ Versus Intrauterine Pressure Catheter (IUPC) in Uterine Contractions Monitoring of Pregnant Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuvo-Group, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP-2000
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Healthy, Pregnant Women

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Study group (Experimental): Healthy 32 weeks or more pregnant women, at an early stage of labor.
  Interventions: Device: INVU™; Device: IUPC; Device: TOCO

INTERVENTIONS:
Device: INVU™ — The subject will undergo continuous recording of the uterine contractions and the fetal heart rate (FHR) for 30 to 60 min using INVU™.
Device: IUPC — The study participants will undergo continuous recording of the uterine contractions by IUPC.
Device: TOCO — Some of the study participants will undergo continuous recording of the uterine contractions and the fetal heart rate (FHR) by TOCO as well.
  Other Names: CTG

SUMMARY:
The primary objective of this research is to assess the agreement between INVU™ and IUPC (the gold standard) during prenatal monitoring of uterine contractions and to assess the safety of INVU™. Additional information comparing INVU™ to TOCO (the standard of care) was also collected.

DETAILED DESCRIPTION:
This multi-center, prospective, comparative, open-label study will be performed in two steps: A training step where up to 40 subjects will be enrolled to confirm uterine contraction performance level.

In the second, validation step, the performance of the uterine contraction detection algorithm will be validated. The validation phase will involve up to 80 subjects.

Sub-study will be implemented in the sites that will monitor the uterine activity of the subjects with TOCO, in addition to INVU™ and IUPC.

Following the screening process, participants subject will undergo continuous recording of the uterine contraction and the fetal heart rate (FHR) for 30 to 60 min using INVU™, Cardiotocograph ((TOCO / CTG), and Intrauterine Pressure Catheters (IUPC). The collected data will be downloaded and comprehensive analysis of the values will be performed offline. Each participant will undergo continuous monitoring by the medical team to identify any safety issue, including but not limited to irritation, sensitization, and potential harmful misuse.

ELIGIBILITY:
Inclusion Criteria:

* Female age between 18-50
* Gestational age ≥32 + 0 weeks
* Singleton gestation
* Ability to understand and sign informed consent
* The subject is within the first stage labor, including early, active and transition phases (cervix is dilated up to 10 cm)
* The subject has an IUPC in place for clinical contraction monitoring
* Exclusion Criteria:
* BMI ≥50 and 15≤ prior pregnancy (Body Mass Index)
* Multiple gestation
* Uncontrolled Hypertension
* Known fetal Anomaly (i.e. major structural)
* Subjects with skin problems in the abdominal area (such as flesh wounds, cuts in the skin, skin rashes, etc.)
* Subjects with implanted electronic devices (pacemaker, defibrillator, etc.)
* Subjects who, in the judgment of the investigator, are likely to be non-compliant or uncooperative during the study
* Subject who is within the second stage labor (cervix is fully dilated to 10 cm or going into the second stage of labor or more)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Study participants are healthy, pregnant women
Enrollment: 80 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the agreement between INVU™ and IUPC (the gold standard) during monitoring of uterine contractions as well as the agreement between Cardiotocography (TOCO) and IUPC, where applicable. | 30-60 minutes per participant
  Three blinded assessors will review the uterine contractions output data (the recordings) from the monitoring devices and determine for each time point whether a contraction occurred. The assessors will not have visibility to the source of the recorded data. Each assessor will review the sessions in a randomized order, while the evaluation will include: a contraction start point, peak, and endpoint. The actual presence of a contraction will be determined by the IUPC.

CONTACTS AND LOCATIONS:
Overall Officials: Nadav Schwartz, MD, Principal Investigator — University of Pennsylvania; Curtis Lowery, MD, Principal Investigator — University of Arkansas
Locations (2):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwartz N, Mhajna M, Moody HL, Zahar Y, Shkolnik K, Reches A, Lowery CL Jr. Novel uterine contraction monitoring to enable remote, self-administered nonstress testing. Am J Obstet Gynecol. 2022 Apr;226(4):554.e1-554.e12. doi: 10.1016/j.ajog.2021.11.018. Epub 2021 Nov 8. PMID 34762863